CLINICAL TRIAL: NCT00940550
Title: A Randomised, Double-Blind, Placebo-Controlled Four-Way Cross-Over Trial to Study the Effects of Prolonged-Release Melatonin, Temazepam and Zolpidem on the Spectral Composition of the EEG During Nocturnal Sleep in Healthy Middle-Aged Men and Women
Brief Title: Study to Investigate the Effects of Melatonin, Temazepam & Zolpidem on Sleep EEG in Men and Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Dr. Malgorzata Knurowska, Surrey Clinical Research Centre
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CRC 266
Record Dates: First submitted 2009-07-15; First posted 2009-07-16 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2009-11

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Temazepam; Zolpidem

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Prolonged-release melatonin 2 mg (Experimental)
  Interventions: Drug: Prolonged-release melatonin
- Temazepam 20 mg (Active Comparator)
  Interventions: Drug: Temazepam
- Zolpidem 10 mg (Active Comparator)
  Interventions: Drug: Zolpidem
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo to match melatonin, zolpidem and temazepam

INTERVENTIONS:
Drug: Prolonged-release melatonin — 2 mg tablet, once.
  Arms: Prolonged-release melatonin 2 mg
Drug: Temazepam — 20 mg capsule, once
  Arms: Temazepam 20 mg
Drug: Zolpidem — 10 mg capsule, once
  Arms: Zolpidem 10 mg
Drug: Placebo to match melatonin, zolpidem and temazepam — Placebo to match melatonin: tablet, once. Placebo to match zolpidem: capsule, once. Placebo to match temazepam: capsule, once.
  Arms: Placebo

SUMMARY:
This study has been designed to compare the effects of melatonin with those of drugs (temazepam and zolpidem) regularly prescribed for the treatment of insomnia, in healthy, middle-aged volunteers.

The study will take place at one centre. Volunteers consenting to participate in the study will have their eligibility confirmed by a screening panel, including spending one night in the sleep clinic to acclimatize to the study procedures. Blood and urine samples will be collected during this overnight visit.

Volunteers continuing to remain eligible will receive, in turn, melatonin, temazepam, zolpidem and placebo as a single dose during 4 treatment phases lasting one night and separated by at least five days. Neither the volunteer nor the study staff will be aware of which drug each volunteer is receiving at each treatment phase.

The volunteer's electrical brain activity will be measured whilst sleeping. Other aspects of sleep, including measures of sleep quality, will also be measured. Urine samples will be collected during each treatment phase.

Volunteers will undergo an assessment of health prior to departure from the clinic at their last treatment phase, and study staff will telephone 2 weeks later to obtain further information on their health status.

The primary study objective is to compare EEG power spectra during nonREM sleep in the slow-wave frequencies following administration with melatonin to temazepam.

DETAILED DESCRIPTION:
This four-way cross-over study has been designed to compare the effects of three drugs used in the treatment of insomnia on the brain electrical activity of healthy middle-aged volunteers during sleep. During each of four treatment phases, volunteers will receive either prolonged-release melatonin, temazepam, zolpidem or placebo, in sequence as governed by a pre-determined randomisation schedule.

The study will be conducted at a single centre clinical research facility (Surrey CRC).

Volunteers who are eligible following screening will be invited to return to the sleep clinic so that they may undergo a one-night period of acclimatisation to the study procedures (the polysomnography [PSG] screen, Visit 2). Following confirmation that the participant has adhered to the protocols restrictions, including tests for drugs of abuse and alcohol use, vital signs will be measured and the actigraph will be replaced. Twice before going to sleep and once on awakening, participants will complete a Karolinska Sleepiness Scale and undergo a Karolinska Drowsiness Test. Participants will then undergo polysomnography, a series of recordings of brain activity using electroencephalography and patterns of breathing, for an eight hour period of sleep. In the evening a cannula will be fitted so that repeat blood samples can be taken and this will be removed the next morning. During the course of the evening three urine samples and four blood samples will be taken for the purpose of assay for melatonin. Three additional blood samples will be taken during the night and urine will be collected. On awakening, urine will be collected and the participant's stability will be assessed using the Romberg test and the Heel-to-Toe Gait test.

Following the PSG screen, volunteers will then undergo four periods of study (Visits 3 through 6), each of one night and separated by at least five days, during which time participants will be administered either a single dose of prolonged-release melatonin or a matching placebo, and a single dose of temazepam, zolpidem or a matching placebo. During each of these periods, the same assessments as those conducted during the PSG screen will be repeated except that blood samples will not be drawn for melatonin assay.

Prior to departure from the sleep centre on each participant's last treatment period (or at withdrawal if earlier), a physical examination including measurement of vital signs will be performed, 12-lead ECG recorded and the clinical safety laboratory evaluations repeated.

Adverse events and concomitant medications will be recorded throughout the study from the time of screening to discontinuation.

Two weeks after the final treatment period, participants will be contacted by telephone to confirm whether they have experienced any adverse events since completion of the study.

A person's melatonin profile is widely recognised as a reliable marker of that individual's timing of the circadian clock. Study participants' plasma melatonin profiles will be measured during the PSG visit. Urinary melatonin will be measured during the PSG visit and all treatment periods.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is able to read and understand the Informed Consent Form (ICF), and understand study procedures.
2. The subject has signed the ICF.
3. Healthy male or female subjects aged 55-64 years inclusive. Attempts will be made to achieve an equal gender ratio through appropriate screening procedures, but a failure to do so will not preclude analysis of the final data set.
4. The subject has a history of the following sleep characteristics during the past three months or more at Visit 1:

   * Bedtime between 22:00-00:00h on at least five nights per week
   * Reported typical nightly sleep duration between 6.5 and 8.5 h
   * The subject has a regular sleep-wake cycle and maintains a regular sleep-wake cycle during the study
5. The subject is a non-smoker who has not used nicotine or nicotine-containing products for at least approximately 6 months. Subjects who have discontinued smoking or the use of nicotine/nicotine containing products for at least approximately 3 months may be enrolled in the study at the discretion of the investigator.
6. The subject is, in the opinion of the investigator, healthy on the basis of a physical examination, medical history, vital signs, ECG, and the results of routine laboratory tests.

Exclusion Criteria:

1. The subject is female AND of childbearing potential. Female volunteers will be considered not of child-bearing potential if they are:

   1. Pre-menopausal women who have been surgically sterilized by bilateral oopherectomy and/or hysterectomy, OR
   2. Post-menopausal, defined as:

      * No spontaneous menstruation for at least one year prior to the first dose,
      * Follicular stimulation hormone (FSH) >18mIU/mL, AND
      * Not lactating.
2. The subject has a known sensitivity to temazepam, zolpidem or melatonin or a history of any allergy that in the opinion of the investigator would contraindicate subject participation.
3. The subject has a BMI of less than 19, or more than 33kg/m or a total body weight of less than 50 kilograms at pre-study (screening) visit. BMI is calculated by taking the subject's weight in kg and dividing by the subject's height in metres, squared.
4. The subject has a score of >5 points on the Pittsburgh Sleep Quality Index (PSQI) scale.
5. The subject has a history of clinically significant sleep pathology according to DSM-IV TRTM or presents symptoms of clinically significant sleep pathology at PSG screening. AHI of >10 and PLMAI of >10.
6. The subject is a shift worker or maintains an irregular sleep-wake schedule during 1 month preceding the screening visit, or travelled within the last month preceding the screening visit and/or during the study to a time zone more than 2 hours different to the current time zone in Surrey.
7. The subject consumes more than three (men) or two (women) units of alcohol per day on average over the 1 month preceding Visit 1(screening visit) [NOTE: 1 unit is equivalent to a half-pint (220mL) of beer or 1 (25mL) measure of spirits or 1 glass (125mL) of wine].
8. The subject consumes more than 5 caffeine-containing beverages per day.
9. Clinically significant psychiatric, cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological (particularly myasthenia gravis), immunological, or haematological disease or abnormality, as determined by the study physician.
10. History of alcohol, narcotic, benzodiazepine, or other substance abuse or dependence within the 12 months preceding Visit 1.
11. Positive urine drug screen at any visit at Surrey CRC (i.e., amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, or opiates). A repeat test will not be allowed.
12. Positive alcohol breath test at any visit to Surrey CRC. A repeat test will not be allowed. [NOTE: subjects must be told to avoid consumption of alcoholic beverages for at least 24 hours prior to attending the Centre].
13. Use of any psychotropic medications such as benzodiazepines, barbiturates and narcotics, or other medications, including over the counter (OTC) and herbal products including melatonin that may affect sleep/wake function, within the 3 months or 5 half-lives preceding Visit 1, whichever is longer, or a need to use any of these medications during the study.
14. Use of any other medication which may interfere with study outcome and/or interfere with IMP within the 2 weeks or 5 half lives preceding Visit 2, with the exception of non-steroidal analgesics, and paracetamol. [NOTE: Concomitant medications which do not influence study outcome and/or do not interfere with IMP may be allowed at the discretion of the investigator].
15. Hereditary problems of galactose intolerance, the Lapp lactase deficiency, or glucose-galactose malabsorption.
16. Currently participating in another clinical trial with an investigational or non-investigational drug or device, or has participated in another clinical trial within the 3 months preceding Visit 1 (screening visit).
17. Concomitant use of HRT by female volunteer.
18. Any condition that, in the investigator's opinion, compromises the volunteer's ability to meet protocol requirements or to complete the study.
19. Subject must be able to refrain from strenuous or unaccustomed exercise such as weight lifting, running and bicycling 24 hours before visits 2, 3, 4, 5 and 6, and 24 hours after visits 2, 3, 4, 5, and 6.

Ages: 55 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
EEG Power density in slow wave frequencies during NREM sleep | Treatment Periods 1 to 4

SECONDARY OUTCOMES:
EEG power density 0.25-32.0 Hz in NREM and REM sleep. EEG power density in the theta frequencies during the Karolinska Drowsiness Test. Objective polysomnography measures of sleep | Treatment Periods 1 to 4

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Daryl Bendel, MBChB, Study Director — Surrey CRC; Dr. Malgorzata Knurowska, MD, Principal Investigator — Surrey CRC; Professor Derk-Jan Dijk, Ph.D., B.S., M.S, Study Chair — Surrey Sleep Research Centre
Locations (1):
- Surrey CRC, University of Surrey, Egerton Road, Guildford, Surrey, United Kingdom